CLINICAL TRIAL: NCT00517491
Title: A Pilot Study to Evaluate the Correlation Between Plasma Lanreotide Levels and GH/IGF-1 Dynamics and Clinical Improvement in Patients With Acromegaly Treated With Lanreotide Autogel (Somatuline ATG)
Brief Title: Study to Evaluate Patients With Acromegaly Treated With Lanreotide Autogel (Somatuline ATG)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative reasons
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-38-52030-725
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — lanreotide

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: lanreotide (Autogel formulation)

INTERVENTIONS:
Drug: lanreotide (Autogel formulation) — 120 mg administered every 28 days via deep subcutaneous injection. A total of 4 injections will be administered during the study.

SUMMARY:
The purpose of the protocol is to evaluate the correlation between plasma lanreotide levels and Growth Hormone (GH)/Insulin Like Growth Factor 1 (IGF-1) dynamics and clinical improvement in patients with acromegaly treated with lanreotide Autogel (Somatuline ATG)

ELIGIBILITY:
Inclusion Criteria:

* Patient on treatment with octreotide LAR 20 mg administered every 28 days for at least 3 months prior to visit 1.
* Patient must have serum GH level ≤ 2.5 ng/mL and serum IGF-1 ≤ 1.3 ULN, 28 days after their last injection of octreotide LAR 20 mg at visit 1.
* Patients must have serum GH level > 2.5 ng/mL AND serum IGF-1 level > 1.3 ULN, 6 or 8 weeks after their last injection of octreotide LAR 20 mg.

Exclusion Criteria:

* The patient has received pituitary radiation therapy of any kind at any time prior to visit 1.
* The patient has received pituitary surgery within 3 months prior to visit 1.
* The patient's serum creatinine is higher than 150 µmol/l.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
GH (basal and during Oral Glucose Tolerance Test (OGTT)) and IGF-1 levels, in acromegalic patients previously treated with octreotide long acting release (LAR) 20 mg. | Weeks 16, 18 & 20
Acromegaly symptoms. | Weeks 16, 18 & 20
Indices of insulin secretion & sensitivity | Weeks 16, 18 & 20
Adverse events | Throughout study

SECONDARY OUTCOMES:
Number of patients with GH levels ≤ 2.5 ng/mL and the number of patients with IGF-1 level < upper limit of normal (ULN). | Weeks 16, 18 & 20.
Serum lanreotide Autogel 120 mg concentrations. | Weeks 16, 18 & 20.
ECG and gallbladder ultrasound | Week 20

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Centro Médico Nacional Siglo XXI, IMSS, Mexico City, Mexico